CLINICAL TRIAL: NCT02353234
Title: Bioavailability of Phenolic Compounds in Wholegrain Bread Compared With White Bread Enriched With Aleurone Fraction
Brief Title: Bioavailability of Phenolic Compounds in Bread
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Parma (Other)
Responsible Party: Principal Investigator, Daniele Del Rio, Associate Professor, University of Parma
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: DDR-001
Record Dates: First submitted 2015-01-27; First posted 2015-02-02 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Dietary Modification
Keywords: Phenolics; Aleurone; Bioavailability; Pharmacokinetics
MeSH Terms: interventions — Bread

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- WHOLEGRAIN BREAD (Active Comparator): Subjects feed with wholegrain bread, for which ferulic acid content has been quantified.
  Interventions: Other: Bread
- WHITE BREAD WITH ALEURONE - 4 (Active Comparator): Subjects feed with white bread with aleurone fraction in the same portion as wholegrain bread.
  Interventions: Other: Bread
- WHITE BREAD WITH ALEURONE - 8 (Active Comparator): Subjects feed with white bread with aleurone fraction, which contains the same quantity of ferulic acid as wholegrain bread.
  Interventions: Other: Bread

INTERVENTIONS:
Other: Bread — In each arm subjects consume bread

SUMMARY:
The consumption of wholemeal cereals has been associated with the reduction of several chronic diseases. The mechanisms behind these protective effects may be linked, besides dietary fiber and micronutrients, to an increased intake of phenolic compounds, mainly, hydroxycinnamates contained in the bran. Among bran fractions, aleurone usually contains the highest concentration of ferulic acid, principally contained as monomeric form and diferulic acid esters linked to arabinoxylans, representing the most relevant subclasses. The aim of the study was to evaluate the absorption of hydroxycinnamates by measuring the urinary excretion of phenolic metabolites in humans fed with two different kind of a commercial bread, as wholegrain bread and a white bread enriched with aleurone fraction. Moreover, the pharmacokinetics of the main phenolic compounds was also evaluated by measuring the circulating metabolites in plasma samples.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18-25 kg/m2

Exclusion Criteria:

* Pregnancy and breastfeeding
* diagnosis of celiac disease
* diagnosed methabolic diseases (diabetes and disorders of glycaemic control, hypertension, dyslipidemia)
* sustained use of nutritional supplements of vitamins, in particular E and C, at the recruitment step
* chronic pharmacological therapy
* antibiotic therapy during the last 40 days

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2014-12; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Phenolic compound bioavailability in wholegrain bread compared with bread enriched with aleurone fraction (urine samples will be filtered and diluted and phenolic compound metabolites will be identified) | 0h; 0-3h; 3-6h; 6-10h; 10-14h; 14-24h; 24-28h; 28-34h; 34-48h.
  Volunteers will collect urine before consuming bread (T0) and for 48 hours after the consumption of the meal test, in each study arms. Urine samples will be collected and stored at -80°C until uHPLC/MS analysis. Prior analysis, urine samples will be filtered and diluted and phenolic compound metabolites will be identified.
  Expected Metabolites:
  Coumaric acid, Hydroxyphenylpropionic acid, Dihydroxyphenylacetic acid, Hippuric acid, Enterolactone, Enterodiol, Coumaric acid sulphate, Phenylpropionic acid sulphate, Vanillic acid sulphate, Hydroxyphenylpropionic acid sulphate, Ferulic acid sulphate, Dihydroferulic acid sulphate, Hydroxyphenylpropionic acid glucuronide, Ferulic acid glucuronide, Enterolactone sulphate, Enterodiol sulphate, Enterolactone glucuronide, Enterodiol glucuronide.

SECONDARY OUTCOMES:
Phenolic compound pharmacokinetics in wholegrain bread compared with bread enriched with aleurone fraction (metabolites identified in Plasma samples that will be collected prior (T0) and after bread consumption in each study arms.) | 0h; 0.5h; 1h; 2h; 4h; 7h; 24h.
  Plasma samples will be collected prior (T0) and after bread consumption in each study arms.
  Expected Metabolites:
  Coumaric acid, Hydroxyphenylpropionic acid, Dihydroxyphenylacetic acid, Hippuric acid, Enterolactone, Enterodiol, Coumaric acid sulphate, Phenylpropionic acid sulphate, Vanillic acid sulphate, Hydroxyphenylpropionic acid sulphate, Ferulic acid sulphate, Dihydroferulic acid sulphate, Hydroxyphenylpropionic acid glucuronide, Ferulic acid glucuronide, Enterolactone sulphate, Enterodiol sulphate, Enterolactone glucuronide, Enterodiol glucuronide.

CONTACTS AND LOCATIONS:
Overall Officials: Daniele Del Rio, Professor, Principal Investigator — University of Parma
Locations (1):
- University of Parma - Department of Food Science, Parma, Italy

REFERENCES:
- [Background] Anson NM, Selinheimo E, Havenaar R, Aura AM, Mattila I, Lehtinen P, Bast A, Poutanen K, Haenen GR. Bioprocessing of wheat bran improves in vitro bioaccessibility and colonic metabolism of phenolic compounds. J Agric Food Chem. 2009 Jul 22;57(14):6148-55. doi: 10.1021/jf900492h. PMID 19537710
- [Background] Del Rio D, Rodriguez-Mateos A, Spencer JP, Tognolini M, Borges G, Crozier A. Dietary (poly)phenolics in human health: structures, bioavailability, and evidence of protective effects against chronic diseases. Antioxid Redox Signal. 2013 May 10;18(14):1818-92. doi: 10.1089/ars.2012.4581. Epub 2012 Aug 27. PMID 22794138
- [Background] Gabrielsson J, Weiner D. Non-compartmental analysis. Methods Mol Biol. 2012;929:377-89. doi: 10.1007/978-1-62703-050-2_16. PMID 23007438
- [Background] Kikuzaki H, Hisamoto M, Hirose K, Akiyama K, Taniguchi H. Antioxidant properties of ferulic acid and its related compounds. J Agric Food Chem. 2002 Mar 27;50(7):2161-8. doi: 10.1021/jf011348w. PMID 11902973
- [Background] Calani L, Ounnas F, Salen P, Demeilliers C, Bresciani L, Scazzina F, Brighenti F, Melegari C, Crozier A, de Lorgeril M, Del Rio D. Bioavailability and metabolism of hydroxycinnamates in rats fed with durum wheat aleurone fractions. Food Funct. 2014 Aug;5(8):1738-46. doi: 10.1039/c4fo00328d. PMID 24977665
- [Background] Luceri C, Giannini L, Lodovici M, Antonucci E, Abbate R, Masini E, Dolara P. p-Coumaric acid, a common dietary phenol, inhibits platelet activity in vitro and in vivo. Br J Nutr. 2007 Mar;97(3):458-63. doi: 10.1017/S0007114507657882. PMID 17313706
- [Background] Mateo Anson N, Hemery YM, Bast A, Haenen GR. Optimizing the bioactive potential of wheat bran by processing. Food Funct. 2012 Apr;3(4):362-75. doi: 10.1039/c2fo10241b. Epub 2012 Feb 15. No abstract available. PMID 22336890
- [Background] Stalmach A, Mullen W, Barron D, Uchida K, Yokota T, Cavin C, Steiling H, Williamson G, Crozier A. Metabolite profiling of hydroxycinnamate derivatives in plasma and urine after the ingestion of coffee by humans: identification of biomarkers of coffee consumption. Drug Metab Dispos. 2009 Aug;37(8):1749-58. doi: 10.1124/dmd.109.028019. Epub 2009 May 21. PMID 19460943
- [Background] Stalmach A, Steiling H, Williamson G, Crozier A. Bioavailability of chlorogenic acids following acute ingestion of coffee by humans with an ileostomy. Arch Biochem Biophys. 2010 Sep 1;501(1):98-105. doi: 10.1016/j.abb.2010.03.005. Epub 2010 Mar 11. PMID 20226754
- [Background] Truswell AS. Cereal grains and coronary heart disease. Eur J Clin Nutr. 2002 Jan;56(1):1-14. doi: 10.1038/sj.ejcn.1601283. PMID 11840174
- [Background] Zaupa M, Scazzina F, Dall'Asta M, Calani L, Del Rio D, Bianchi MA, Melegari C, De Albertis P, Tribuzio G, Pellegrini N, Brighenti F. In vitro bioaccessibility of phenolics and vitamins from durum wheat aleurone fractions. J Agric Food Chem. 2014 Feb 19;62(7):1543-9. doi: 10.1021/jf404522a. Epub 2014 Feb 6. PMID 24450764